CLINICAL TRIAL: NCT05372055
Title: Malignant Pleural Effusions: Evaluating the psYchosocial Impact of Indwelling Pleural Catheters on Patients (MY-IPC)
Brief Title: Malignant Pleural Effusions: Evaluating the psYchosocial Impact of Indwelling Pleural Catheters on Patients
Acronym: MY-IPC
Status: Completed | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 313971
Record Dates: First submitted 2022-05-09; First posted 2022-05-12 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-03

CONDITIONS: Malignant Pleural Effusion; Indwelling Pleural Catheter
Keywords: Malignant Pleural Effusion; Indwelling Pleural Catheter; Psychosocial
MeSH Terms: conditions — Pleural Effusion, Malignant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Indwelling Pleural Catheter: Patients with malignant pleural effusions managed by IPC insertion as per standard of care
  Interventions: Other: Semi-structure interviews

INTERVENTIONS:
Other: Semi-structure interviews — Semi-structured interview focusing on psychosocial impact of living with an IPC to be performed at 2 weeks and 6-8 weeks post IPC insertion

SUMMARY:
The purpose of this study is to better understand the impact that Indwelling Pleural Catheters have on patients with malignant pleural effusions from a psychosocial point of view.

DETAILED DESCRIPTION:
After being informed about the study, all patients giving written informed consent will undergo a baseline assessment including disease and social characteristics on the day of their Indwelling Pleural Catheter (IPC) insertion. At 2 weeks and 6-8 weeks post insertion, they will be contacted via telephone for a semi-structured interview focusing on the psychosocial impact that the IPC has had on their lives. Data surrounding the medical care of the IPC will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study
* Aged 18 years or above
* Diagnosis of malignant pleural effusion
* Will be undergoing IPC insertion for management of their malignant pleural effusion
* Have the means to be contacted and be able to conduct an interview in English via telephone within the study timeframe

Exclusion Criteria:

* Inability to consent
* Estimated life expectancy of <4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with symptomatic malignant pleural effusions treated with indwelling pleural catheter insertion
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2023-05-08 (Actual); Study Completion 2023-05-08 (Actual)

PRIMARY OUTCOMES:
The psychosocial impact of living with an indwelling pleural catheter in patients with malignant pleural effusions | 2 weeks
  Qualitative data
The psychosocial impact of living with an indwelling pleural catheter in patients with malignant pleural effusions | 6-8 weeks
  Qualitative data

SECONDARY OUTCOMES:
Links between psychosocial impact experienced by patients and their baseline, disease or social characteristics | 2 weeks and 6-8 weeks
  Qualitative data
Links between psychosocial impact experienced by patients and their IPC care characteristics | 2 weeks and 6-8 weeks
  Qualitative data

CONTACTS AND LOCATIONS:
Overall Officials: Parthipan Sivakumar, BM,BSc, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- Guy's & St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American Thoracic Society. Management of malignant pleural effusions. Am J Respir Crit Care Med. 2000 Nov;162(5):1987-2001. doi: 10.1164/ajrccm.162.5.ats8-00. No abstract available. PMID 11069845
- [Background] Roberts ME, Neville E, Berrisford RG, Antunes G, Ali NJ; BTS Pleural Disease Guideline Group. Management of a malignant pleural effusion: British Thoracic Society Pleural Disease Guideline 2010. Thorax. 2010 Aug;65 Suppl 2:ii32-40. doi: 10.1136/thx.2010.136994. No abstract available. PMID 20696691
- [Background] Feller-Kopman DJ, Reddy CB, DeCamp MM, Diekemper RL, Gould MK, Henry T, Iyer NP, Lee YCG, Lewis SZ, Maskell NA, Rahman NM, Sterman DH, Wahidi MM, Balekian AA. Management of Malignant Pleural Effusions. An Official ATS/STS/STR Clinical Practice Guideline. Am J Respir Crit Care Med. 2018 Oct 1;198(7):839-849. doi: 10.1164/rccm.201807-1415ST. PMID 30272503
- [Background] Bibby AC, Dorn P, Psallidas I, Porcel JM, Janssen J, Froudarakis M, Subotic D, Astoul P, Licht P, Schmid R, Scherpereel A, Rahman NM, Maskell NA, Cardillo G. ERS/EACTS statement on the management of malignant pleural effusions. Eur J Cardiothorac Surg. 2019 Jan 1;55(1):116-132. doi: 10.1093/ejcts/ezy258. PMID 30060030
- [Background] Ayaz-Alkaya S. Overview of psychosocial problems in individuals with stoma: A review of literature. Int Wound J. 2019 Feb;16(1):243-249. doi: 10.1111/iwj.13018. Epub 2018 Nov 4. PMID 30392194
- [Background] Michálková H. PSYCHOSOCIAL PROBLEMS OF STOMA CLIENTS. :9.
- [Background] Di Gesaro A. The psychological aspects of having a stoma: a literature review. Gastrointestinal Nursing. 2016 Mar 2;14(2):38-44.
- [Background] Moller T, Adamsen L. Hematologic patients' clinical and psychosocial experiences with implanted long-term central venous catheter: self-management versus professionally controlled care. Cancer Nurs. 2010 Nov-Dec;33(6):426-35. doi: 10.1097/NCC.0b013e3181dc1908. PMID 20562617
- [Background] Stern JM, Jacyna N, Lloyd DA. Review article: psychological aspects of home parenteral nutrition, abnormal illness behaviour and risk of self-harm in patients with central venous catheters. Aliment Pharmacol Ther. 2008 May;27(10):910-8. doi: 10.1111/j.1365-2036.2008.03646.x. Epub 2008 Feb 12. PMID 18284646
- [Background] Davies HE, Mishra EK, Kahan BC, Wrightson JM, Stanton AE, Guhan A, Davies CW, Grayez J, Harrison R, Prasad A, Crosthwaite N, Lee YC, Davies RJ, Miller RF, Rahman NM. Effect of an indwelling pleural catheter vs chest tube and talc pleurodesis for relieving dyspnea in patients with malignant pleural effusion: the TIME2 randomized controlled trial. JAMA. 2012 Jun 13;307(22):2383-9. doi: 10.1001/jama.2012.5535. PMID 22610520
- [Background] Thomas R, Fysh ETH, Smith NA, Lee P, Kwan BCH, Yap E, Horwood FC, Piccolo F, Lam DCL, Garske LA, Shrestha R, Kosky C, Read CA, Murray K, Lee YCG. Effect of an Indwelling Pleural Catheter vs Talc Pleurodesis on Hospitalization Days in Patients With Malignant Pleural Effusion: The AMPLE Randomized Clinical Trial. JAMA. 2017 Nov 21;318(19):1903-1912. doi: 10.1001/jama.2017.17426. PMID 29164255
- [Background] Muruganandan S, Azzopardi M, Fitzgerald DB, Shrestha R, Kwan BCH, Lam DCL, De Chaneet CC, Rashid Ali MRS, Yap E, Tobin CL, Garske LA, Nguyen PT, Stanley C, Popowicz ND, Kosky C, Thomas R, Read CA, Budgeon CA, Feller-Kopman D, Maskell NA, Murray K, Lee YCG. Aggressive versus symptom-guided drainage of malignant pleural effusion via indwelling pleural catheters (AMPLE-2): an open-label randomised trial. Lancet Respir Med. 2018 Sep;6(9):671-680. doi: 10.1016/S2213-2600(18)30288-1. Epub 2018 Jul 20. PMID 30037711
- [Background] Bhatnagar R, Keenan EK, Morley AJ, Kahan BC, Stanton AE, Haris M, Harrison RN, Mustafa RA, Bishop LJ, Ahmed L, West A, Holme J, Evison M, Munavvar M, Sivasothy P, Herre J, Cooper D, Roberts M, Guhan A, Hooper C, Walters J, Saba TS, Chakrabarti B, Gunatilake S, Psallidas I, Walker SP, Bibby AC, Smith S, Stadon LJ, Zahan-Evans NJ, Lee YCG, Harvey JE, Rahman NM, Miller RF, Maskell NA. Outpatient Talc Administration by Indwelling Pleural Catheter for Malignant Effusion. N Engl J Med. 2018 Apr 5;378(14):1313-1322. doi: 10.1056/NEJMoa1716883. PMID 29617585
- [Background] Prieto L, Thorsen H, Juul K. Development and validation of a quality of life questionnaire for patients with colostomy or ileostomy. Health Qual Life Outcomes. 2005 Oct 12;3:62. doi: 10.1186/1477-7525-3-62. PMID 16219109
- [Background] Maslow AH. Motivation and personality. New York: Harper & Row; 1970.
- [Background] Kiger ME, Varpio L. Thematic analysis of qualitative data: AMEE Guide No. 131. Med Teach. 2020 Aug;42(8):846-854. doi: 10.1080/0142159X.2020.1755030. Epub 2020 May 1. PMID 32356468
- [Background] Braun V, Clarke V. Using thematic analysis in psychology. Qualitative Research in Psychology. 2006 Jan 1;3:77-101.
- [Background] Rehman KU, Liang J, Sivakumar P. P103 Provision of pleural disease care in the pandemic era: A single centre experience. Thorax. 2021 Nov 1;76(Suppl 2):A123-A123.
- [Derived] Zhang J, Liang J, Agoramoorthy L, Montalvo S, Kadwani O, Radcliffe G, Sivakumar P. Psychosocial impact of living with an indwelling pleural catheter in patients with malignant pleural effusions: a thematic analysis. BMJ Open Respir Res. 2025 Jul 8;12(1):e002993. doi: 10.1136/bmjresp-2024-002993. PMID 40628689